CLINICAL TRIAL: NCT03838705
Title: The Relationship Between Postoperative Oxygenation and STOP-BANG Questionnaire and 4-V Tool in Preoperative Bariatric Surgery Patients
Brief Title: The Relationship Between Postoperative Oxygenation and STOP-BANG Questionnaire and 4-V Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Collaborators: Sibel Ocak Serin (Unknown); Aysun Isiklar (Unknown)
Responsible Party: Principal Investigator, Gulsah Karaoren, Associate professor, Umraniye Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SS1
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hypoxia; Bariatric Surgery
Keywords: stop-bang, bariatric surgery, obesity, hypoxia
MeSH Terms: conditions — Hypoxia; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bariatric surgery patients (Other): patients aged 18-65 years with ASA status II-III, BMI>40 who were undergoing bariatric surgery operation
  Interventions: Procedure: hypoxia; Procedure: normooxy

INTERVENTIONS:
Procedure: hypoxia — It was accepted that hypoxia developed in patients with SpO2< 92 or falling over 20% compared to preoperative values.
Procedure: normooxy — It was accepted that patients with SpO2 between 100-92 mmHg

SUMMARY:
In our study, we aimed to investigate the relationship between STOP-BANG and 4-Variable Screening questionnaires in postoperative period in patients who underwent bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40
* bariatric surgery patients

Exclusion Criteria:

* malignancy
* patients who are unable to complete the questionnaire
* patients who needs laparotomy

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
SpO2 | 48 hours
  Peripheral Oxygen Saturation

SECONDARY OUTCOMES:
STOP-BANG | preoperative 24 hours
  The value of STOP-BANG questionnaire
4-V Tool | preoperative 24 hours
  The value of 4-V Tool

CONTACTS AND LOCATIONS:
Overall Officials: Sibel O Serin, MD, Study Director — Umraniye Research Hospital
Locations (1):
- Istanbul Umraniye Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No